CLINICAL TRIAL: NCT06330818
Title: IMAGINE - Imaging in Moyamoya Disease
Brief Title: Imaging in Moyamoya Disease - Study to Investigate Different Imaging Technologies for a Better Understanding of Various Imaging Techniques to Evaluate Cerebral Hemodynamics, Disease-activity and Possibly the Etiology in Moyamoya Patients
Acronym: IMAGINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMAGINE Moyamoya; 528291394 (Other Grant/Funding Number: German Research Council (DFG))
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-03

CONDITIONS: Moyamoya Disease; Moyamoya
Keywords: Stroke; Moyamoya; EC-IC Bypass
MeSH Terms: conditions — Moyamoya Disease; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moyamoya patients (Experimental): Newly diagnosed Moyamoya patients who will follow a standardized imaging and biosampling protocol. Possible surgical or conservative treatment will not be influenced by this study.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: H2 15O PET/CT; Other: Biosampling
- Control group (No Intervention): Healthy patients and patients with intracerebral atherosclerotic disease are used as comparators for the results of biosampling.

INTERVENTIONS:
Diagnostic Test: MRI — Patients will get special MRI sequences (CO2-triggered BOLD MRI, Vessel-wall imaging, resting state BOLD MRI) to identify cerebral vasoreactivity and disease activity.
  Arms: Moyamoya patients
Diagnostic Test: H2 15O PET/CT — Patients will get H2 15O PET/CT with acetazolamide challenge to define the cerebral vasoreserve for comparison with fMRI Images
  Arms: Moyamoya patients
Other: Biosampling — Patients do get a venous puncture for blood analysis on circulating endothelial cells and virus PCR analysis
  Arms: Moyamoya patients

SUMMARY:
Aim of this study is to improve patient care in Moyamoya Patients by improving Imaging technologies and aiming to identify factors involved in disease progression.

Main tasks are:

* Analysis of CO2-triggered BOLD fMRI for analysis of cerebral hemodynamics in comparison to H2 15O PET/CT
* Analysis of longitudinal changes of contrast enhancement in vessel-wall imaging and correlation of disease activity with biosampling
* Definition of a standardized recommendation for pre- and postoperative imaging of Moyamoya patients

DETAILED DESCRIPTION:
Moyamoya Disease (MMD) is a rare disease defined by a bilateral stenosis or occlusion of the terminal internal carotid artery (ICA) and proximal arteries of the circle of willis. The stenosis is usually accompanied by fine collateral vessels appearing as "a puff of smoke" on conventional DSA giving the disease its name (Japanese). The disease is known to progress over time in 20-40% of adult patients, also to initially not affected vessels. To prevent from ischemic or hemorrhagic strokes, most patients need microsurgical revascularization with extracranial-intracranial (EC-IC) bypasses for the affected cerebrovascular territories. The indication for a possible revascularization should always be decided based on functional imaging identifying cerebrovascular territories with an insufficient reserve capacity. The "gold-standard" for measuring the cerebrovascular reserve is H2 15O PET/CT with Acetazolamide challenge (ACZ), whereat also SPECT and different MRI techniques are used but with less sensitivity. Main drawback of H2 15O PET/CT is its very limited availability, high costs, the need to inject ACZ and radiation exposure. Further, the costs of H2 15O PET/CT for Moyamoya patients are not covered by the German health insurance system as no valid high-quality studies are available to prove a possible benefit of this examination.

Throughout the last years the investigators have focused our research on different MRI techniques in Moyamoya patients aiming to find reliable examinations for the evaluation of the cerebral blood flow and to detect and monitor disease progression:

The investigators' newly developed semi-automated algorithms for the evaluation of CO2-triggered BOLD MRI (breathhold fMRI) sequences to identify a reduced vasoreactivity showed a promisingly high correlation to the results of the cerebrovascular reserve measurements as seen in PET/CT. Further, the investigators were able to show that disease progression can be predicted by a temporary contrast enhancement of the vessel wall seen over approximately 24 months as high-resolution vessel-wall imaging was performed consequently in all patients.

Therefore, the main goals of this study are to improve patient care in Moyamoya patients with the following three key elements:

1. Defining the value of CO2 triggered BOLD MRI in the evaluation of cerebral hemodynamics pre- and postoperatively compared to H2 15O PET/CT aiming to possibly prove or reduce the need for PET/CT examinations.
2. Understanding radiographic and pathophysiologic processes causing disease progression as seen by vessel-wall imaging to enable timely revascularization or possibly non-surgical treatment of this disease in the future.
3. Possible new insights in disease-pathophysiology and progression as seen in vessel wall imaging by correlating imaging results with biosampling (peripheral blood
4. Defining a standardized recommendation for pre- and postoperative hemodynamic and MR-morphologic evaluation of Moyamoya patients based on the results of this study.

As secondary objectives the following elements will be analyzed:

1. Neuropsychological impairment in correlation to the hemodynamic and MR-morphologic status of the brain.
2. Feasibility of resting-state fMRI to evaluate cerebral vasoreactivity.

To achieve these goals, the investigators are planning to prospectively include 50 Moyamoya patients in this study with a standardized imaging, neuropsychological testing and biosampling protocol with a two-year follow-up. Under the assumption of a homogenous inclusion of patients, recruitment should be finished after two years with one year of follow-up after the inclusion of the last patient. This cohort will provide reliable information on standardized diagnostic patterns and possibly a broader understanding of pathophysiology causing disease development and progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of Moyamoya Disease
* Patients able to understand the study and to give their informed consent

Exclusion Criteria:

* Cerebral vascular disease caused by atherosclerosis
* Vasculitis
* Contraindications to MRI
* Contraindications to PET/CT
* Pregnancy
* Inability to give informed consent
* Renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Value of CO2-triggered BOLD MRI compared to PET/CT | From enrollment until maximum of 24 months
  Analysis of comparability of fMRI-based vasoreactivity and PET/CT based vasoreserve (Signal change in percent)

SECONDARY OUTCOMES:
Vessel-Wall contrast enhancement | From enrollment until maximum of 24 months
  Analysis of vessel-wall contrast enhancement as predictor for disease-activity (Intensity of contrast enhancement relative to reference tissue on MRI)
Circulating endothelial cells | From enrollment to a maximum of 24 months
  FACS-based analysis of circulating endothelial cells as indicator for disease activity (absolute number of respective circulating endothelial cells subgroup)
PCR-based virus sampling | From enrollment until maximum 24 months
  Analysis of possible virus infections as indicator for disease etiology (absolute number of Virus DNA based on PCR results)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Neurosurgery, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available anonymized upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR